CLINICAL TRIAL: NCT05061992
Title: A Trial to Improve Quality of Life in People With Cirrhosis - the Michigan Kristalose Trial
Brief Title: A Trial to Improve Quality of Life in People With Cirrhosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elliot B. Tapper, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00204056
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Cirrhosis
Keywords: Hepatic Encephalopathy; Liver Disease; Cirrhosis and portal hypertension
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Liver Diseases; Hypertension, Portal | interventions — Lactulose

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactulose (Experimental)
  Interventions: Drug: Lactulose
- No treatment (No Intervention): Subjects will complete baseline and outcome assessments at 28 days and no intervention or placebo will be prescribed.

INTERVENTIONS:
Drug: Lactulose — Participants will take 20 grams (dissolved in 4ounces of water/beverage) doses of lactulose twice daily (upon awakening and then 4 hours later) for 28 days.
  In addition, outcome measurements will be completed at baseline and day 28.
  Other Names: Kristalose
  Arms: Lactulose

SUMMARY:
This trial is being completed to evaluate whether a crystallized form of lactulose (Kristalose) will improve quality of life, sleep and cognitive function in patients with cirrhosis that have not been diagnosed with Hepatic Encephalopathy (HE), but report reduced quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis - must meet one of the following criteria:

  1. liver biopsy, OR
  2. history of cirrhosis complication: ascites, variceal bleeding, hepatic encephalopathy, OR
  3. 2 of the following 4 criteria:

     1. Ultrasound, Computed tomography (CT) or Magnetic resonance imaging (MRI) findings of cirrhosis (cirrhotic appearing liver, splenomegaly, varices, ascites)
     2. Fibroscan liver stiffness score >13 Kilopascal (kPa)
     3. Laboratory testing: aspartate aminotransferase (AST)/platelet ratio index (APRI) >2.0
     4. CT, MRI or Esophagogastroduodenoscopy (EGD) showing presence of esophageal varices

        Exclusion Criteria:
* Non-English speaking
* Pregnancy (self-reported)
* Unable or unwilling to provide consent
* History of liver transplant
* Disorientation at the time of enrollment, Dementia, or Treated Memory Disorder
* History of prior lactulose use or HE within 6 months
* Metastatic solid malignancy or blood malignancy
* Hemoglobin A1C > 12 (within past year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Tapper, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactulose | No Treatment
Started | 28 | 28
Completed | 25 | 27
Not Completed | 3 | 1
Not completed — Excess bowel movements | 1 | 0
Not completed — Complications of Medical Care | 1 | 0
Not completed — Diarrhea Prior to Starting Therapy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactulose | No Treatment | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (11.9) | 61.8 (11.3) | 60.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 28 | 56
Short Form-8 Health Survey (SF-8) [Mean (Standard Deviation); unit: score on a scale] — 0 (lowest quality of living) to 100 (highest quality of living)
  score on a scale | 57.2 (18.3) | 61.1 (17.0) | 59.2 (17.7)
Animal Naming Test [Mean (Standard Deviation); unit: Count of Animals Named] — Number of unique animals named within 1 minute by the participant.
  Count of Animals Named | 17.9 (5.3) | 18.3 (6.5) | 18.1 (5.8)
Sleep Quality [Mean (Standard Deviation); unit: Score on a Scale] — Overall sleep quality was measured on a 5-point Likert scale, with a range of 1 (very bad sleep quality) to 5 (very good sleep quality).
  Score on a Scale | 2.5 (0.8) | 2.5 (0.8) | 2.5 (0.8)
Activity Impairment [Mean (Standard Deviation); unit: Score on a Scale] — Single survey question where participants responded on a Likert scale of 0 (no impairment) to 10 (complete impairment)
  Score on a Scale | 5.4 (1.9) | 5.7 (2.1) | 5.6 (2.1)
Participants Who Fell in Past 90 Days [Count of Participants; unit: Participants] — Yes or no question on whether participant had experienced at least 1 fall in the past 90 days.
  Participants | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Short Form-8 Health Survey (SF-8) at 28 Days
Description: The SF-8 is an abbreviated version of an original 36-item health survey (SF-36). It is a generic, multipurpose, quality of life instrument, containing psychometrically based physical and mental health summary measures. The eight domains are general health, physical functioning, role physical, bodily pain, vitality, social functioning, mental health, and role emotional. Scores from the domains are combined and range from 0 (lowest quality of living) to 100 (highest quality of living).
Time Frame: 28 days
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lactulose | No Treatment
Number analyzed (Participants) | 25 | 27
score on a scale
  Change in SF-8 from Baseline | 8.1 [3.7 to 12.4] | 6.55 [2.3 to 10.8]
  End of Trial SF-8 | 70.9 [63.9 to 77.9] | 63.84 [57.1 to 70.6]
Statistical Analysis 1: Comparison: Lactulose vs No Treatment; Change in SF-8; Test type: Superiority; p = 0.6, ANCOVA
Statistical Analysis 2: Comparison: Lactulose vs No Treatment; End of trial SF-8; Test type: Superiority; p = 0.2, ANCOVA

2. Secondary Outcome: Animal Naming Test (ANT)
Description: Number of unique animals named within 1 minute by the participant. Values below show the change from baseline and the results from the test taken 28 days later.
Time Frame: 28 days
Measure: Mean (95% Confidence Interval); unit: Count of Animals Named
Arm/Group | Lactulose | No Treatment
Number analyzed (Participants) | 25 | 27
Count of Animals Named
  Change in ANT | 3.7 [2.1 to 5.4] | -0.15 [-1.7 to 1.4]
  End of trial ANT | 21.2 [18.9 to 23.6] | 18.52 [16.3 to 20.8]
Statistical Analysis 1: Comparison: Lactulose vs No Treatment; Change in ANT; Test type: Superiority; p = 0.001, ANCOVA
Statistical Analysis 2: Comparison: Lactulose vs No Treatment; End of trial ANT; Test type: Superiority; p = 0.09, t-test, 2 sided

3. Secondary Outcome: Change in Overall Sleep Quality
Description: Overall sleep quality was measured on a 5-point Likert scale, with a range of 1 (very bad sleep quality) to 5 (very good sleep quality).
Time Frame: Change between baseline (day 0) and 28 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lactulose | No Treatment
Number analyzed (Participants) | 25 | 27
score on a scale | 0.4 [0.1 to 0.7] | 0.0 [-0.3 to 0.3]
Statistical Analysis 1: Comparison: Lactulose vs No Treatment; Test type: Superiority; p = 0.05, ANCOVA

4. Secondary Outcome: Regular Daily Activity Impairment
Description: Single-question survey given to participants at baseline and again 28 days later. Participants ranked their daily activity impairment on a Likert scale of 0 (no impairment) to 10 (complete impairment)
Time Frame: 28 days
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lactulose | No Treatment
Number analyzed (Participants) | 25 | 27
score on a scale | 3.0 [1.9 to 4.0] | 4.8 [3.8 to 5.8]
Statistical Analysis 1: Comparison: Lactulose vs No Treatment; Test type: Superiority; p = 0.02, ANCOVA

5. Secondary Outcome: Participants Who Fell
Description: Yes or no question on whether participant had experienced at least 1 fall in the past 28 days.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lactulose | No Treatment
Number analyzed (Participants) | 25 | 27
Participants | 1 | 3
Statistical Analysis 1: Comparison: Lactulose vs No Treatment; Test type: Superiority; p = 0.6, Fisher Exact

6. Secondary Outcome: Daily Bowel Movements
Description: Results show the percentage of days in a 28-day span in which participants experienced more than 5 daily bowel movements. All participants analyzed in each arm were included in calculating the results using the following formula: (days with >5 bowel movements) / (patient-days in study) The results are presented as a single number because they are a point estimate of a population level proportion
Time Frame: 28 days
Measure: Number; unit: % of participant-days with >5 bowels
Arm/Group | Lactulose | No Treatment
Number analyzed (Participants) | 25 | 27
% of participant-days with >5 bowels | 5 | 2
Statistical Analysis 1: Comparison: Lactulose vs No Treatment; Test type: Superiority; p = 0.2, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Lactulose | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/28
Other Adverse Events (participants affected / at risk) | 1/28 | 3/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lactulose (N=28) | No Treatment (N=28)
Complications from Liver Disease (Hepatobiliary disorders) | 1 | 1 — Hospitalizations occurred for participants because of complications with pre-existing liver disease.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lactulose (N=28) | No Treatment (N=28)
Fall (Musculoskeletal and connective tissue disorders) | 1 | 3 — Non-injurious fall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT05061992/Prot_SAP_000.pdf